CLINICAL TRIAL: NCT04430517
Title: Effects of Orally Administered Nicotinamide Riboside on Bioenergetic Metabolism, Oxidative Stress and Cognition in Mild Cognitive Impairment and Mild Alzheimer's Dementia
Brief Title: Effects of Nicotinamide Riboside on Bioenergetics and Oxidative Stress in Mild Cognitive Impairment/Alzheimer's Dementia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Fei Du, Director, Laboratory for High-Field Imaging and Translational Neuroscience, Mclean Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2020P001652; 1R01AG066670 (NIH)
Record Dates: First submitted 2020-05-29; First posted 2020-06-12 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-09

CONDITIONS: Mild Cognitive Impairment; Mild Alzheimer Disease
Keywords: Mild Cognitive Impairment; Bioenergetics; Mild Alzheimer's Dementia
MeSH Terms: conditions — Cognitive Dysfunction | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Mild Cognitive Impairment and Alzheimer's Dementia (Experimental): Participants will take 4 pills every day, each containing 250 mg NR (NIAGEN® by Chromadex; www.chromadex.com), via the oral route, for 12 weeks.
  Interventions: Drug: Nicotinamide riboside

INTERVENTIONS:
Drug: Nicotinamide riboside — Participants will take 4 pills every day, each containing 250 mg NR (NIAGEN® by Chromadex; www.chromadex.com), via the oral route, for 12 weeks.
  Other Names: Chromadex NIAGEN

SUMMARY:
The primary aim of this study is to investigate the effects of exogenously administered nicotinamide riboside (NR) on brain energy metabolism, oxidative stress, and cognitive function in individuals with mild cognitive impairment (MCI) and mild Alzheimer's dementia (AD).

DETAILED DESCRIPTION:
Mitochondrial function is mediated, in part, by nicotinamide adenine dinucleotide (NAD). Unfortunately, decreases in NAD+ levels are associated with normal aging, and also with numerous diseases such as AD. Accumulating evidence suggests that NR can enhance mitochondrial function and help slow or reverse these age-related abnormalities. Numerous preclinical and clinical studies have been performed using NR and related compounds to boost NAD+ level in human subjects with various diseases or animal models. However, no studies to date have investigated in vivo metabolic and bioenergetic changes (target engagement) associated with NR supplementation. In this project, we aim to investigate the neurobiological mechanisms and clinical effects of NR in patients with MCI and mild AD using in vivo novel neuroimaging techniques.

ELIGIBILITY:
Inclusion Criteria:

* Ability of the participant and/or his/her legally authorized representative to understand the purpose and risks of the study, to provide signed and dated informed consent, and to authorize the use of confidential health information.
* Ability to speak and read fluently in English
* 55-89 years old (inclusive)
* Normal or corrected to normal hearing and vision
* Meet clinical diagnostic criteria for MCI or Mild AD, according to the following criteria:

  1. CDR Global Score of 0.5 (MCI) or 1.0 (mild AD)
  2. 2018 NIA-AA guidelines for MCI/mild AD
* Study partner available for the duration of trial participation
* At least one copy of the APOE ε4 allele or AD+ including Amyloid positive PET scan, Tau positive PET Scan (MK6240 et al.), or CSF AD biomarkers [i.e., amyloid-beta beta (Aβ42) total (T)-tau, and phosphorylated (P)-tau]
* An aggregate risk score > 4 according to the risk analysis method developed by Sabbagh et al. (2017)
* For individuals who are taking niacin (or a vitamin supplement with niacin) of >200mg, the completion of a two-week wash-out period

Exclusion Criteria:

* Current serious or unstable medical or neurological condition that could affect cognitive functioning, as determined by study clinician
* Clinically unstable mood or anxiety disorder within 6 months prior to screening, as determined by study clinician
* Lifetime history of psychotic disorder (i.e. Schizophrenia, Schizoaffective Disorder), as determined by study clinician
* Diagnosis of a mitochondrial disorder
* Any MRI safety contraindications
* History of drug hypersensitivity or intolerance to NR
* Transient ischemic attack or stroke within 1 year prior to screening
* History of alcohol or substance abuse within prior year, as determined by study clinician and urine toxicology screen
* History of head injury rated as moderate or worse, per DSM-5 criteria
* History of seizure within prior 10 years
* Current use of medication with known adverse effects on cognition (benzodiazepines, barbiturates, opiate analgesics, first generation antipsychotic medication, centrally acting anticholinergics, sedating antihistamines, tricyclic anti-depressants)
* Change in dose of any psychiatric medications within 4 weeks of screening visit
* Prior use of L-DOPA, any anti-Parkinsonian medication, or prior treatment with anti-amyloid immunotherapy
* Current use of putative mitochondrial enhancers and antioxidants (e.g carnitine, creatine Co-Q10, N-acetyl cysteine [NAC], pramipexole)
* Initiation of treatment or change in dosing of acetylcholinesterase inhibitors (AChEIs) and memantine within 4 weeks of baseline visit
* Prior use of prescription narcotics 4 weeks before baseline visit
* Female subjects who are pregnant or breastfeeding
* The use of current use of niacin (or a vitamin supplement with niacin) >200mg within the last two weeks prior to study visit.
* Current or lifetime history of cancer.

Ages: 55 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-03-02 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Changes in brain NAD+ | Baseline, 6 and 12 weeks, pre- and post- 1000 mg NR daily
  Changes in brain NAD+ levels
Changes in brain redox state | Baseline, 6 and 12 weeks, pre- and post- 1000 mg NR daily
  Changes in brain NAD+/NADH ratio

SECONDARY OUTCOMES:
Changes in mitochondrial function | Baseline, 6 and 12 weeks, pre- and post- 1000 mg NR daily
  Changes in brain CK/ATPase activity
Changes in antioxidant glutathione (GSH) levels | Baseline, 6 and 12 weeks, pre- and post- 1000 mg NR daily
  Changes in brain GSH levels

OTHER OUTCOMES:
Changes in cognitive status | Baseline, 6 and 12 weeks, pre- and post- 1000 mg NR daily
  Changes in Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) scores. The RBANS provides a total score from 40-160, with a higher score indicating a better outcome.
Changes in functional status | Baseline, 6 and 12 weeks, pre- and post- 1000 mg NR daily
  Changes in Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL) scores. The ADCS-ADL provides a total score from 0-78, with a higher score indicating lower severity and a better outcome.
Changes in mood | Baseline, 6 and 12 weeks, pre- and post- 1000 mg NR daily
  Changes in Patient Health Questionnaire (PHQ-9) scores. The PHQ-9 provides a total score from 0-27, with a higher score indicating more symptoms of depression.
Changes in behavioral or psychiatric symptoms resulting from memory problem | Baseline, 6 and 12 weeks, pre- and post- 1000 mg NR daily
  Changes in The Neuropsychiatric Inventory Questionnaire (NPI-Q) responses. The NPI-Q is scored in 12 domains which assess the severity and distress of specific mood, behavioral, or psychiatric symptoms resulting from memory problems. Higher scores indicate greater severity or caregiver distress associated with each of the behavioral and psychiatric symptoms.
Changes in spirituality and religious beliefs | Baseline and 12 weeks, pre- and post- 1000 mg NR daily
  Changes in responses to series of brief psychometrically valid and reliable measures of spirituality/religion administered in order to evaluate spiritual/religious predictors of adjustment to AD as indexed by emotional, behavioral, neurocognitive, and neural assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Fei Du, PhD, Principal Investigator — Mclean Hospital; Brent Forester, MD, MSc, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The proposed research will include data and biosamples from 50 subjects who will receive open-label treatment with nicotinamide riboside (NR) throughout the duration of the 12-week study. At the time of publication of the primary results or within 9 months of database lock, whichever comes first, we will create deidentified datasets, which could be available for research purposes to qualified individuals within the scientific community.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: At the time of publication of the primary results or within 9 months of database lock, whichever comes first, we will create deidentified datasets, which could be available for research purposes to qualified individuals within the scientific community.
Access Criteria: Data are available to users only under a data-sharing agreement. All users will provide to PIs a proposal of hypotheses, variables needed to test these hypotheses, and plans for dissemination of findings. All users will indicate in a signed document: (1) a commitment to using the data only for research purposes and not to identify any participant, clinician, or plan; (2) a plan for securing the data using appropriate technology/data use protocols; (3) an agreement to either destroy or return the data once analyses are completed or by a specific negotiated date; (4) appropriate IRB approval; (5) a commitment that the information provided to users will not be used for commercial purposes, will not be redistributed to third parties, or shared with any others not on the research team; (6) adequate funding/resources to analyze the data and publish results. All findings generated will be described via peer-reviewed articles in scientific journals made available via PubMed Central.